CLINICAL TRIAL: NCT04689009
Title: Multi-centre, Randomized Controlled, Prospective Study on the Speed of Healing, Life Quality and Cost-effectiveness of the Treatment With the Blue Light Medical Device EmoLED vs a Standard Treatment for Leg Ulcers (L.U.C.E. Study)
Brief Title: Leg Ulcers Standards of Care Enhancement
Acronym: LUCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emoled (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EmoLED_003
Record Dates: First submitted 2020-11-18; First posted 2020-12-30 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Venous Leg Ulcer; Mixed Leg Ulcer
Keywords: leg ulcer; photobiomodulation; blue light; wound healing
MeSH Terms: conditions — Varicose Ulcer; Leg Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOC Group (Active Comparator): SOC Group (or control group) will follow the standard therapy with visits twice a week. More specifically, the treatment consists of: dressing change, cleansing and eventual debridement of the lesion, the topic treatment and compression bandage.
  Interventions: Procedure: current Standards Of Care
- EmoLED Group (Experimental): EmoLED Group will be visited once a week. Therapy in this case includes, in addition to the standard therapy, a treatment with EmoLED device; it consists in irradiating each 5 cm diameter area of the lesion for 60 seconds, with the blue light emitted by the device. For lesions larger than 5 cm, several applications will be applied on adjacent areas, until the whole lesion is covered.
  Interventions: Device: EmoLED; Procedure: current Standards Of Care

INTERVENTIONS:
Device: EmoLED — The treatment with EmoLED, in addition to the SOC, will be performed during each visit for 60 seconds on each 5 cm diameter sub-area of the selected lesion.
  Arms: EmoLED Group
Procedure: current Standards Of Care — The lesions will be cleansed with saline solution and, if necessary, surgical debridement will be performed with the most suitable method. At this point, if patient is included in EmoLED Group, the EmoLED treatment starts. After EmoLED application (EmoLED Group) or after cleansing (SOC Group), a polyurethane foam dressing will be applied on the lesion. In case of clinical signs of infection, a silver dressing will be applied.
  Then an elasto-compressive double layer dressing of the limb with cohesive fixation bielastic latex-free bandage will be carried out.

SUMMARY:
Multi-center, prospective,randomized controlled study on the speed of healing, life quality and cost-effectiveness of the treatment with a blue light medical device (EmoLED) versus existing Standards Of Care (SOC) for patients with leg ulcers.

The aim of LUCE - "Leg Ulcers Standards of Care Enhancement" clinical trial is to verify the clinical efficacy of a portable battery-powered device blue LEDs based. This study aims to compare the existing SOC (consisting in two visits per week) to a protocol that requires only one visit per week, during which the EmoLED treatment is administered in addition to the current therapy.

It is expected to register a difference in efficacy between EmoLED Group and SOC Group, in terms of "healing rate", intended as a reduction of the wound area, but also as a progress, in a broad sense, of the overall clinical situation of the lesion, in terms of pain and quality of life.

-Endpoint- The primary endpoint is the comparison of the outcomes in terms of healing rate of lesions treated with SOC (SOC Group) versus lesions treated with EmoLED (EmoLED Group), on week 16th.

Patients 80 patients will be recruited (40 patients per group), following these inclusion/exclusion criteria:

Inclusion criteria:

* Subjects suffering from venous and mixed skin ulcers;
* Presence of a lesion < 100 cm² of area and < 1 cm in depth;
* Men and women ≥ 18 years old;
* The patient must be able to understand the aims of the clinical trial and provide informed consent in writing;
* Chronicity of the lesion: at least 8 weeks.

Exclusion criteria:

* Patients who participated in clinical trials about skin ulcers healing during the previous month;
* Patients who are not able to understand the aims of the trial;
* Patients with pressure ulcers;
* Patients with diabetic foot ulcers;
* Patients with circumferential leg ulcer (due to the difficulties in analysing the pictures);
* Patients with clearly infected ulcers or with systemic infection;
* Patients with ulcers caused by critical ischemia;
* Patients with a self-harm past that can purposely alter the process of healing;
* Patients with psychiatric disorders;
* Pregnancy or breast feeding;
* Patients with neoplasms or other diseases involving the use of cytostatic or immunosuppressive drugs;
* Patients with limited lifespan;
* Patients with photosensitizing illnesses or that take photosensitizing drugs. All inclusion and exclusion criteria must be satisfied before recruitment. Any concomitant phar-macological therapy must be maintained.

-Medical and surgical procedures- The lesions will be cleansed with saline solution and, if necessary, surgical debridement will be performed with the most suitable method. At this point, if patient is included in EmoLED Group, the EmoLED treatment starts. After EmoLED application (EmoLED Group) or after cleansing (SOC Group), a polyurethane foam dressing will be applied on the lesion. In case of clinical signs of infection, a silver dressing will be applied.

Then an elasto-compressive double layer dressing of the limb with cohesive fixation bielastic la-tex-free bandage will be carried out.

The treatment with EmoLED, in addition to the SOC, will be performed during each visit for 60 seconds on each 5 cm diameter sub-area of the selected lesion.

In case of multiple lesions matching with both inclusion and exclusion criteria, they will be all treated following the same protocol, depending on the group to which the patient belongs; in this case the Principal Investigator will fill out a data-collection form and take pictures just of the le-sion with the wider area.

-Follow up procedure- The patient is called upon to go to the follow-up check after 4 weeks from the healing or, other-wise, from the end of the trial (16 weeks). The follow-up visit will be used to confirm the occurred healing and verify the absence of relapses and/or undesirable effects (if the wound appeared completely healed) or to value the healing progress for the unhealed lesions.

DETAILED DESCRIPTION:
EmoLED is CE marked as a phototherapy device for the treatment of skin lesions. It is intended for use by medical personnel in a hospital or outpatient setting. The patients' demographic consists of individuals with skin lesions that are at least 16 old, regardless of their ethnicity. EmoLED is conceived and designed to treat chronic and acute lesions of the skin by healthcare professionals such as doctors and nurses; in particular the EmoLED treatment is part of the wound bed preparation.

EmoLED treatment is additional to the conventional therapy consisting in the lesions cleansing and dressing with conventional or advanced medications.

The blue light emitted by the device interacts with the endogenous chromophores of the skin triggering reactions that lead to the activation of certain cellular pathways. In particular, the wavelength emitted by the device is absorbed by Protoporphyrin IX present in Cytochrome C, an essential protein for cellular respiration at the mitochondrial level. The energy absorbed is used by the cell to increase the production of ATP, a fundamental molecule for all the processes involved in tissue repair. In addition, blue light is able to stimulate the production of ROS (Reactive Oxygen Species) through the excitation of flavins and flavoproteines. Nowadays, multiple evidence has been produced about how ROS can be considered signal transducers of numerous cellular pathways. This consideration validates the evidence that ROS (at physiological concentrations) are crucial for multiple cellular functions such as differentiation, proliferation, migration and contraction.

A way through which EmoLED can act in tissue repair is the chain of mitochondrial electronic transport. EmoLED in particular can act on the last two complexes that contain Cytochrome C, that is sensitive to visible light in the range of emission of the device.

The resulting effect is the strengthening of this process and the increase in ATP production, related to the development of a proton gradient dependent on the electron transport chain. The increase of ATP production determines an increment of the available energy for the cell that can intensify its metabolic activity, a necessary process during the repair of an injury that involves activation of different cell types and an additional energy effort for the organism.

The device has been designed and set to deliver a power density of about 7 J/cm2 in an acceptable treatment time for both doctor and patient: 60 seconds for each circular area of 5 cm diameter that needs to be treated. The choice of the duration of the treatment was also made on the basis of what is stated in literature on thermal damage: the treatment induces a temperature between 45 and 50ºC in the treated area, ideal condition to stimulate the reversible and physiological phenomena that are wanted.

Ethical considerations:

The study will be submitted to the Ethical Committee of each investigator hospital for approval and in any case will be performed according to the GCP, the Helsinki Declaration and the Italian laws and requirements in the matter of human clinical trials.

Informed consent procedure:

The Principal Investigator (PI) or their delegate selects the enrolled patients on the basis of the inclusion and exclusion criteria of the study. Once the patient's correspondence with the study's criteria has been verified, the PI or their delegate asks the patient for consent to use the EmoLED treatment device, and briefly explains the characteristics of the device, the expected effect, the possible trial-related risks, the guarantees to protect the confidentiality of the collected information. The PI asks the patient if they are interested in participating, leaving them twenty-four hours to decide. If the patient manifests their interest to participate in the study, during their next visit they will sign the Informed Consent and will decide whether to inform their family doctor of their participation in the study. The patient must give their availability to return to the structure every week for the trial observation time, including the follow up visit.

A copy of the Informed Consent, subscribed by the patient and by the Principal Investigator and a copy of the study information will be given to the patients.

Measurable parameters:

The key data and lesion's pictures of each patient will be collected in the Data Collection Form, following the enrollment and the signing of the Informed Consent:

* SOC Group: (32 treatments are planned during 16 weeks, 2 times per week)
* EmoLED Group: (16 treatments are planned during 16 weeks, 1 time per week)

The parameters used to define the study result will be based on:

* Photographic images of lesions treated with EmoLED and control lesions
* Data Collection Form filled by the medical staff during the visit
* Economic-organizational impact survey
* Survey on the usability of the device (SUS)
* Detection of pain through VAS scale

Registration of clinical data:

The parameters of the Data Collection Form are acquired on paper, and conserved in both paper and digital form; the pictures of the lesion are acquired and kept in digital form.

During each visit, a picture of the lesion will be taken so that the process of healing can be valued also in a visual way.Each picture will be named with the patient code and the date of the visit. In case of multiple lesions matching with both inclusion and exclusion criteria, they will be all treated following the same protocol, depending on the group of treatment, but only the lesion with the wider area will be registered; to distinguish the area of interest, the perilesional tissue will be labelled with single-use permanent markers.

Data Collection Form:

The Data Collection Form is unique for each patient and includes: Clinical Section, Quality Life Section and Economic Section. The Clinical Section contains identification code of the patient, date of birth, sex, etiology of the ulcer, any eventual concurrent disease, any drug therapy (in terms of active substances), ulcer's date of onset, date of entry to the facility.

The second part of the form is organized as a matrix where the row represents the measurable parameters for each time of observation (reported in column).

The investigator marks with an "X" the chosen value for each parameter and the most suitable description. The Principal Investigator will also fill a check list, for each visit, to ensure that also the pain level has been measured and that the picture of the lesion has been taken.

There is also a "Notes" section to register information not planned at first, that might be helpful during the data analysis.

The last part of the Data Collection Form is about follow-up visit. The Data Collection Form is already completed with the patient's recruitment code and the group they belong to, so that the allocation to the EmoLED Group and the SOC Group is random. The allocation sequence of the group is generated by Matlab.

On each visit, the patient will be asked to rate their current pain level (VAS scale 0-10).

The quality section survey will be administered on the first and last visits, and also every 4 weeks. In detail, standard questionnaires as the EQ-5D2 and the Wound-Qol3 will be administered, both available and validated in Italian language.

Specific questionnaires for recognition of costs (Economic section) will be administered to patients and their primary caregiver (if present) during the first visit, with the aim of identifying the resources absorbed by the patients (and their caregivers) treated in the two different approaches. The consumption of resources will be measured by gathering information about the quantification of direct health costs (visits, hospitalizations, emergency healthcare, medications etc…), direct non-health-related costs (informal medical assistance, transportation and accommodation costs for each visit etc..) and indirect costs (productivity loss for both the patient and the caregiver/s) and also by taking into account both the costs associated with the adherence to the treatment, taking the first visit as a reference parameter, and the costs related to complications and events associated with the ulcer that determined the need for treatments/ exams and/or medical evaluations. The Principal Investigator will be given also a questionnaire to determine the costs incurred by their facility for handling patients with leg ulcers.

The questionnaires meant to value customer satisfaction, complexity and helpfulness of EmoLED device will be administered to doctors and to healthcare personnel involved in the treatment at the end of the trial.

Image Acquisition:

For the 16 weeks of the trial, during each visit a picture of the lesion will be taken, so that the process of healing can be valued also in a visual way. Each picture will be named with the patient code and the date of the visit. The quantitative analysis about the size of the lesions through the collected pictures will be performed at certain time points: at the beginning, in the middle and at the end of the treatment.

The image analysis is made through an appropriate analysis algorithm that measures the area of the lesion (mm²). The lesion must be fully and frontally framed to obtain an optimal analysis.The ruler with patient's ID code and date must appear in every picture. It is important that the ruler is placed straight and in-focus to have the scale reference. If there is a wide lesion that needs more than one picture it's advisable to locate several markers around the lesion and take photos of adjacent areas, including at least two visible markers of the previous picture, to have the complete image of the lesion through a sequential photo array.

Bias:

The staff participating in the study is trained on the correct use of the device and accessories, as well as on the correct execution of the clinical protocol and on the compilation of the related forms. In any case, the EMOLED staff is always available to the team for any clarification or doubt during the study.

In order to promote a more homogeneous operation between the various centres, joint training sessions are organized and documents which serve as guidelines for the most critical passages or the ones which require particular attention, such as recording, saving and transmitting data, are prepared.

In order to avoid bias during the procedure of allocation in groups of patients enrolled in the study, it should be noted that the randomization grid is not distributed to the investigators: instead, paper folders are distributed containing the data collection forms. The progressive patient ID is on the outside of the folders, while on the inside a label is placed with the assignment of the patient to one of the two groups (SOC or EmoLED treatment), which reflects the randomization grid. These folders are closed through an adhesive label with the signature of the Head of Clinical Affairs of the sponsoring company.

Patients selection:

All patients that satisfy all the inclusion criteria, both hospitalised and outpatient, will be considered for inclusion in this study.

It will be used a standard procedure to value patients that includes the anamnesis evaluation and a physical examination. A total of 80 subjects will be recruited, 40 per arm at the facilities involved in the clinical study. Each one of the four sites involved will enroll 20 patients.Since this is a multicentric investigation with competitive recruitment the number of patients per site can vary, depending on the recruitment capability of each site.

Once the patient has signed the informed consent, the Principal Investigator enters the data in the Enrollment Registry, checking all the inclusion and exclusion criteria; if all criteria are met, the patient is considered to be enrolled in the clinical study.

Known or predictable factors that may impair outcomes and interpretation of outcomes:

A different therapy standard between participating centers and/or within the same center can lead to very variable outcomes between one patient and another, all other conditions being equal. This problem is tackled by indicating in detail the therapy to be followed depending on the type of lesion.

An incorrect recording of photographic images does not make it possible to determine the area of the lesion via software. This problem is tackled by providing precise instructions on the correct use of the tools available for the retrieval of images.

Discontinuity of patients can affect recovery times. Before recruiting a patient, the doctor ensures that the patient is available to go, with the required timing, to the clinic, for the scheduled visits. This fact is underlined several times when providing study information to the patient.

Interruption and withdrawal of subjects from the clinical trial:

Patients who miss the visits for two consecutive weeks, before/until the 14th week, and the patients who miss the visits for one week, after the 14th week, will be reached by phone by the Principal Investigator to assess their availability to go on with the study; in the event that the patient does not intend to continue with the visits at the centre, they will be excluded from the study.Also, the patient who will turn out to be absent for more than half of the sessions will be excluded as well.

Following the resignation or withdrawal from the study by a patient, their data collection form will be identified, scanned and archived.

If a patient withdraws from the study, the PI or his delegate records the event in the Patient Identification Register and on the Data Collection Form and stores all documentation.

Monitoring plan of the clinical investigation:

To guarantee the conformity with ICH/GCP guidelines, the Clinical Research Coordinator (CRC) will be responsible for the study to be carried out in full observance of the Standard Operating Procedures, of the Protocol and other written instructions.

The main responsibilities of the CRC are to ensure adherence to the Protocol, to make sure that the data are accurately and fully registered and reported and to verify that the Informed Consent was obtained and registered for each subject before the beginning of the study.

The CRC will keep in touch and meet the Principal Investigator on a regular basis throughout the whole duration of the study. The CRC will be allowed to check the various documents (Data Collection Forms, CRF and other related documents containing original data) related to the study in order to verify the conformity with the Protocol and to ensure the accuracy of recorded data.

Quality assurance, control procedures, data management and record-keeping:

All the information gathered during the Study will be considered strictly confidential. The patients' consent to the registration of personal data will be requested at the time of recruitment; nevertheless the data collection forms will contain the Identification Code of the patient and their date of birth only. In order to guarantee the correct traceability of all parties involved, the number of the Study and the naming of the Center will be included as well.

At the end of the Study, all data will be archived using the appropriate safety measures at the Coordinating Site for a minimum of ten years.

If a patient withdraws their consent to data processing, they will be immediately destroyed to ensure total confidentiality, in addition each investigator will keep a copy of the study's documentation for at least two years after its conclusion.

The Principal Investigator builds and is responsible for the updating and custody of the Patient Identification Register or Enrollment Register.

The Patient Identification Register includes personal data of patients who agreed to take part in the study, the identification number assigned to the patient, their illness, indication of the eventual exclusion from the recruitment with its justification and date of recruitment.The patient code is constituted by a three-digit number: the first one indicates the center's number, as stated in this protocol, and the other two are sequential numbers, starting from 01. Only the PI and, at their discretion, the members of their team have knowledge of the identities of patients enrolled in the study.

Adverse Events:

Despite all the information in our possession and physical characteristics and performances of the device that do not suggest the possible occurrence of and adverse event, it is taken into consideration the possibility that said event could take place.

The morbid condition of each patient will be monitored the whole time of the study. During each visit any sign manifested by the patient will be carefully observed; in fact, the subject will be encouraged to report any symptom with direct questions, such as: "How have you been feeling since our last visit?". They will also be prompted to spontaneously report any adverse events that occurred during the study.

Any significant clinical anomaly encountered over the course of the study will be monitored and observed until its normalisation, or until it will be clinically explainable.

If during the procedure an unfavourable eventuality is reported, it shall be considered as an Adverse Event, if Serious Adverse Event or not it will be decided according to customary criteria.

Safety follow-up for subjects:

* The subjects that withdrew from the experimentation after the treatment with the device under study for any reason,
* The subjects who present Adverse Events up until thirty days from the last visit or the last follow-up check (whichever of the two eventualities is the latter),
* All the subject who still present Adverse Events upon completion of the study will be monitored until the test results are not back to baseline, or is no longer expected from them to change, or until the investigator does not determine that those results are no longer clinically relevant.

Statistics- Calculation of the sample size: 80 patients will be recruited during the study; they will be randomized 1:1 to the SOC Group and the EmoLED Group. In the SOC group, which follows the standard treatment, patients will be visited twice a week. The EmoLED Group will undergo medical examination once a week; in this case, therapy will consist in the standard treatment plus EmoLED treatment. This sample size is sufficient to compare the average rate of the injured area reduction, considering Student-T test for the comparison between independent samples, by establishing α = 0.05, power level (1-β) = 0,8, under the assumption to have an area reduction rate after 16 weeks amounting to 50% in SOC Group (control group), a difference of 20% between EmoLED Group (experimental group) and SOC Group, a standard deviation of averages equal to 50% of the mean values and a bilateral hypothesis.

Statistical analysis: The average rate of reduction of the injured area between the two groups will be compared using the Student-T-test, the quality of life in both groups at the baseline, after 16 weeks and the difference with the baseline will be compared using Student-T-test for independent samples. Linear regression models will be used to value the differences between the groups to exclude any confounding factors. Due to the usually asymmetrical nature of cost distribution, the comparison of the costs related to the treatment and control group, in both the NHS and society perspective, will be made using the non-parametric Mann-Whitney U test. Generalized linear regression models will be used to value the differences between the groups to eliminate any confounding factors. The cost-effectiveness of both treatments in the time frame of the study (16 weeks) will be valued by calculating the incremental cost-effectiveness ratio (ICER) and expressed in terms of incremental costs for "quality adjusted years (QALY). Extrapolations of results about the cost-effectiveness that simulate longer time-frames will be made considering decision-making models (e.g. Markov models) and eventually including the data gathered during the study with literary data and/or evidence from other studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects suffering from venous and mixed skin ulcers;
* Presence of a lesion < 100 cm² of area and < 1 cm in depth;
* Men and women ≥ 18 years old;
* The patient must be able to understand the aims of the clinical trial and provide informed consent in writing;
* Chronicity of the lesion: at least 8 weeks.

Exclusion Criteria:

* Patients who participated in clinical trials about skin ulcers healing during the previous month;
* Patients who are not able to understand the aims of the trial;
* Patients with pressure ulcers;
* Patients with diabetic foot ulcers;
* Patients with circumferential leg ulcer (due to the difficulties in analysing the pictures);
* Patients with clearly infected ulcers or with systemic infection;
* Patients with ulcers caused by critical ischemia;
* Patients with a self-harm past that can purposely alter the process of healing;
* Patients with psychiatric disorders;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Romanelli, MD, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana; Stefano Gasperini, MD, Study Director — Medical Advisor
Locations (5):
- Italy (5):
  - Ospedale Briolini, ASST Bergamo EST, Gazzaniga, Bergamo
  - Ospedale Felice Lotti, Pontedera, Pisa
  - Geriatrics Unit, Presidio Ospedaliero di Rete San Bassiano, ULSS 7 Pedemontana, Bassano del Grappa, Vicenza
  - Dermatology Unit AOU Policlinico Sant'Orsola - Malpighi, Bologna
  - Dermatology Unit, Azienda Ospedaliero Universitaria Pisana, Stabilimento di S. Chiara, Pisa

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after publication

REFERENCES:
- [Background] Clark RA. Cutaneous tissue repair: basic biologic considerations. I. J Am Acad Dermatol. 1985 Nov;13(5 Pt 1):701-25. doi: 10.1016/s0190-9622(85)70213-7. PMID 2416789
- [Background] Mast BA, Schultz GS. Interactions of cytokines, growth factors, and proteases in acute and chronic wounds. Wound Repair Regen. 1996 Oct;4(4):411-20. doi: 10.1046/j.1524-475X.1996.40404.x. PMID 17309691
- [Background] Nwomeh BC, Yager DR, Cohen IK. Physiology of the chronic wound. Clin Plast Surg. 1998 Jul;25(3):341-56. PMID 9696897
- [Background] Hackam DJ, Ford HR. Cellular, biochemical, and clinical aspects of wound healing. Surg Infect (Larchmt). 2002;3 Suppl 1:S23-35. doi: 10.1089/sur.2002.3.s1-23. PMID 12573037
- [Background] Calderhead (2007), The photobiological basis behind light-emetting diode (LED) phototherapy, Laser therapy
- [Background] Beani JC, Jeanmougin M. [Narrow-band UVB therapy in psoriasis vulgaris: good practice guideline and recommendations of the French Society of Photodermatology]. Ann Dermatol Venereol. 2010 Jan;137(1):21-31. doi: 10.1016/j.annder.2009.12.004. Epub 2009 Dec 29. French. PMID 20110064
- [Background] Adamskaya N, Dungel P, Mittermayr R, Hartinger J, Feichtinger G, Wassermann K, Redl H, van Griensven M. Light therapy by blue LED improves wound healing in an excision model in rats. Injury. 2011 Sep;42(9):917-21. doi: 10.1016/j.injury.2010.03.023. PMID 22081819
- [Background] Son GY, Hong JH, Chang I, Shin DM. Induction of IL-6 and IL-8 by activation of thermosensitive TRP channels in human PDL cells. Arch Oral Biol. 2015 Apr;60(4):526-32. doi: 10.1016/j.archoralbio.2014.12.014. Epub 2014 Dec 25. PMID 25575297
- [Background] Bertin S, Aoki-Nonaka Y, de Jong PR, Nohara LL, Xu H, Stanwood SR, Srikanth S, Lee J, To K, Abramson L, Yu T, Han T, Touma R, Li X, Gonzalez-Navajas JM, Herdman S, Corr M, Fu G, Dong H, Gwack Y, Franco A, Jefferies WA, Raz E. The ion channel TRPV1 regulates the activation and proinflammatory properties of CD4(+) T cells. Nat Immunol. 2014 Nov;15(11):1055-1063. doi: 10.1038/ni.3009. Epub 2014 Oct 5. PMID 25282159
- [Background] Xu T, Wu BM, Yao HW, Meng XM, Huang C, Ni MM, Li J. Novel insights into TRPM7 function in fibrotic diseases: a potential therapeutic target. J Cell Physiol. 2015 Jun;230(6):1163-9. doi: 10.1002/jcp.24801. PMID 25204892
- [Background] Kleinpenning MM, Smits T, Frunt MH, van Erp PE, van de Kerkhof PC, Gerritsen RM. Clinical and histological effects of blue light on normal skin. Photodermatol Photoimmunol Photomed. 2010 Feb;26(1):16-21. doi: 10.1111/j.1600-0781.2009.00474.x. PMID 20070834
- [Background] Niemz MH (1996), Laser-tissue interactions: fundamentals and applications.
- [Background] Rossi et al. (2010), A blue-LED-based device for selective photocoagulation of superficial abrasions: theoretical modeling and in vivo validation, Photonic Therapeutics and Diagnostics VI, Proceedings of SPIE Volume: 7548.
- [Background] Meaume S, Dissemond J, Addala A, Vanscheidt W, Stucker M, Goerge T, Perceau G, Chahim M, Wicks G, Perez J, Tacca O, Bohbot S. Evaluation of two fibrous wound dressings for the management of leg ulcers: results of a European randomised controlled trial (EARTH RCT). J Wound Care. 2014 Mar;23(3):105-6,108-11, 114-6. doi: 10.12968/jowc.2014.23.3.105. PMID 24633056
- [Background] Hansson C. The effects of cadexomer iodine paste in the treatment of venous leg ulcers compared with hydrocolloid dressing and paraffin gauze dressing. Cadexomer Iodine Study Group. Int J Dermatol. 1998 May;37(5):390-6. doi: 10.1046/j.1365-4362.1998.00415.x. PMID 9620490
- [Background] Marston WA, Carlin RE, Passman MA, Farber MA, Keagy BA. Healing rates and cost efficacy of outpatient compression treatment for leg ulcers associated with venous insufficiency. J Vasc Surg. 1999 Sep;30(3):491-8. doi: 10.1016/s0741-5214(99)70076-5. PMID 10477642
- [Background] F. Petrella, Progetto SIUC (Studio Incidenza Ulcere Cutanee), 1 gennaio 2015 - 31 dicembre 2016, AIUC
- [Background] Vitse J, Bekara F, Byun S, Herlin C, Teot L. A Double-Blind, Placebo-Controlled Randomized Evaluation of the Effect of Low-Level Laser Therapy on Venous Leg Ulcers. Int J Low Extrem Wounds. 2017 Mar;16(1):29-35. doi: 10.1177/1534734617690948. Epub 2017 Feb 17. PMID 28682676

RESULTS

PARTICIPANT FLOW:
Groups:
- SOC Group: SOC Group (or control group) will follow the standard therapy with visits twice a week. More specifically, the treatment consists of: dressing change, cleansing and eventual debridement of the lesion, the topic treatment and compression bandage.
  current Standards Of Care: The lesions will be cleansed with saline solution and, if necessary, surgical debridement will be performed with the most suitable method. At this point, if patient is included in EmoLED Group, the EmoLED treatment starts. After EmoLED application (EmoLED Group) or after cleansing (SOC Group), a polyurethane foam dressing will be applied on the lesion. In case of clinical signs of infection, a silver dressing will be applied.
  Then an elasto-compressive double layer dressing of the limb with cohesive fixation bielastic latex-free bandage will be carried out.
- EmoLED Group: EmoLED Group will be visited once a week. Therapy in this case includes, in addition to the standard therapy, a treatment with EmoLED device; it consists in irradiating each 5 cm diameter area of the lesion for 60 seconds, with the blue light emitted by the device. For lesions larger than 5 cm, several applications will be applied on adjacent areas, until the whole lesion is covered.
  EmoLED: The treatment with EmoLED, in addition to the SOC, will be performed during each visit for 60 seconds on each 5 cm diameter sub-area of the selected lesion.
  current Standards Of Care: The lesions will be cleansed with saline solution and, if necessary, surgical debridement will be performed with the most suitable method. At this point, if patient is included in EmoLED Group, the EmoLED treatment starts. After EmoLED application (EmoLED Group) or after cleansing (SOC Group), a polyurethane foam dressing will be applied on the lesion. In case of clinical signs of infection, a silver dressing will be applied.
  Then an elasto-compressive double layer dressing of the limb with cohesive fixation bielastic latex-free bandage will be carried out.
Period: Overall Study
Arm/Group | SOC Group | EmoLED Group
Started | 41 | 42
Completed | 34 | 37
Not Completed | 7 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SOC Group | EmoLED Group | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 11 | 17
  >=65 years | 35 | 31 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.2 (10.06) | 73.6 (11.83) | 75.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 18 | 18 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 41 | 42 | 83

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change of the Wound Area
Description: It is expected to demonstrate the equivalence between EmoLED Group treatment (consisting in EmoLED treatment + SOC treatment, once a week) and SOC Group treatment (consisting in SOC treatment, twice a week), in terms of percentage change of the wound area, at week 16 and at Follow-up visit (at week 20) from baseline.
  The percentage reduction is measured by calculating: (initial area of the wound - final area of the wound) / initial area of the wound x 100.
Time Frame: Baseline,16 weeks, 20 weeks
Population: Per Protocol population
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | SOC Group | EmoLED Group
Number analyzed (Participants) | 34 | 37
percentage of change
  Area variation at week 16 from baseline | 42.41 (24.58) | 60.75 (26.29)
  Area variation at week 20 from baseline | 25.18 (26.45) | 72.16 (30.59)

2. Secondary Outcome: Healing Time Evaluation
Description: Evaluation of the healing time of the lesions treated with the standard method (SOC Group) versus the lesions treated with the EmoLED (EmoLED Group), through the Data Collection Form, considering the elapsed time between the first visit and the event of interest (the reaching of healing)
Time Frame: 16 weeks
Population: Per Protocol population
Measure: Mean (Standard Error); unit: percent change per week
Arm/Group | SOC Group | EmoLED Group
Number analyzed (Participants) | 34 | 37
percent change per week | 2.16 (0.333) | 3.45 (0.319)

3. Secondary Outcome: Incidence of the Treatment (Standard vs EmoLED Protocol) in Life Quality
Description: Difference of the life quality (QoL) score at 16 week minus the baseline score (week1) assessed by Wound-Qol3 questionnaire (value 0 indicates the best level of quality of life, 4 the worst).
Time Frame: 16 weeks
Population: Patients who filled the first and the last questionnaire
Measure: Mean (Standard Deviation); unit: Score difference
Arm/Group | SOC Group | EmoLED Group
Number analyzed (Participants) | 38 | 35
Score difference | 0.6 (0.7) | 0.7 (0.8)

4. Secondary Outcome: Costs Related Evaluation
Description: Evaluation of costs related to the EmoLED Group and SOC Group, in both the NHS and society perspective, through economic-organizational impact survey. The costs are reported per patient per study period.
Time Frame: 16 weeks
Population: Patients who filled the economic questionnaire
Measure: Mean (Full Range); unit: Euros
Arm/Group | SOC Group | EmoLED Group
Number analyzed (Participants) | 38 | 42
Euros | 7,313 [1,168 to 9,341] | 3,076 [451 to 3,610]

5. Secondary Outcome: Percent Change in VAS Scale Evaluation
Description: Change of perceived pain through VAS scale ("Visual Analog Scale" in which 0 is the minimum value and the better outcome, and 10 is the maximum value and worse outcome) in both groups.
Time Frame: 16 weeks
Population: Per Protocol population
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | SOC Group | EmoLED Group
Number analyzed (Participants) | 25 | 29
percentage change | 65.20 (40.25) | 77.76 (39.72)

6. Secondary Outcome: Satisfaction, Complexity and Helpfulness Evaluation of the Device Assessed by SUS
Description: Evaluation of satisfaction, complexity and helpfulness of EmoLED device, considering both the perspective of patients, and the one of doctors and health care providers involved through a survey on the usability of the device (SUS - System Usability Scale, which includes 10 questions. Participants will classify each question from 1 to 5 based on how much they agree with the statement they are reading. 5 means they agree completely, 1 means they disagree vehemently).
Time Frame: 16 weeks
Population: Healthcare personnel who filled the satisfaction questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale (1 worst - 5 best)
Arm/Group | EmoLED Group
Number analyzed (Participants) | 9
units on a scale (1 worst - 5 best) | 3.96 (0.33)

7. Secondary Outcome: Cost-effectiveness Evaluation
Description: Evaluation of cost-effectiveness using EmoLED in the treatment of ulcers through economic-organizational impact survey. To calculate cost-effectiveness, the cost differential, between EmoLED group and Control group, was evaluated in terms of quality adjusted life years (QALY), obtaining the Incremental Cost-Effectiveness Ratio (ICER).
Time Frame: 16 weeks
Population: Patients who filled the economic questionnaire
Measure: Number; unit: Euro/QALY
Arm/Group | SoC Group | EmoLED Group
Number analyzed (Participants) | 38 | 42
Euro/QALY | 1934.13 | 758.50

ADVERSE EVENTS:
Time Frame: From the time of enrollment to the last visit under the protocol (16 weeks, or less in case of healing)
Arm/Group | SOC Group | EmoLED Group
All-Cause Mortality (participants affected / at risk) | 1/41 | 1/42
Serious Adverse Events (participants affected / at risk) | 2/41 | 1/42
Other Adverse Events (participants affected / at risk) | 1/41 | 1/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOC Group (N=41) | EmoLED Group (N=42)
Erysipelas (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOC Group (N=41) | EmoLED Group (N=42)
Bullous pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythematous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI will not disclose information about the Trial without the consent of the Sponsor. These confidentiality obligations will remain in force until the information is made public by the Promoter. The PI must submit the manuscript to the Promoter, at least 60 days before publication. The Sponsor will then have 45 days to suggest changes to the Investigator.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT04689009/Prot_SAP_001.pdf